CLINICAL TRIAL: NCT03226444
Title: A Double-Masked, Randomized, Multi-Center Phase 2 Study to Evaluate the Efficacy and Safety of Lacripep™ in Subjects With Dry Eye Associated With Primary Sjögren's Syndrome
Brief Title: Lacripep™ in Subjects With Dry Eye Associated With Primary Sjögren's Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TearSolutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LOS-001
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Primary Sjögren Syndrome; Dry Eye
Keywords: Dry Eye; Primary Sjogren's Syndrome; Sjogren's Syndrome
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.005% Lacripep (Experimental): 0.005% Lacripep ophthalmic solution
  Interventions: Drug: 0.005% Lacripep
- 0.01% Lacripep (Experimental): 0.01% Lacripep ophthalmic solution
  Interventions: Drug: 0.01% Lacripep
- placebo (Placebo Comparator): placebo solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.005% Lacripep — One drop (approximately 50 microliters) of 0.005% ophthalmic solution will be administered three times a day (TID) to both eyes for four weeks.
  Arms: 0.005% Lacripep
Drug: 0.01% Lacripep — One drop (approximately 50 microliters) of 0.01% ophthalmic solution will be administered three times a day (TID) to both eyes for four weeks.
  Arms: 0.01% Lacripep
Drug: Placebo — One drop (approximately 50 microliters) of placebo solution will be administered three times a day (TID) to both eyes for four weeks.
  Arms: placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of two strengths of Lacripep™ ophthalmic solution versus placebo administered three times daily for four weeks in subjects with a diagnosis of Dry Eye associated with documented Primary Sjögren's Syndrome

DETAILED DESCRIPTION:
This is a multi-center, randomized, placebo-controlled, double-masked, parallel-group study. Subjects will be randomized into three treatment groups: 0.005%, or 0.01% Lacripep™, or placebo in a 1:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet the following criteria will be selected:

1. Subjects who are age 18 years of age or older at the time of obtaining informed consent.
2. Subjects with a documented prior history or current diagnosis of Primary Sjögren's Syndrome according the American-European Consensus Group Sjögren's Syndrome Criteria (Appendix 4; must meet either 4 out of 6 total criteria OR 3 out of 4 signs). Note: Subjects who are on systemic (oral) therapy for the treatment of Sjögren's Syndrome must be on stable systemic treatment defined as the same treatment for the immediately prior 90 days.
3. Subjects with a history of dry eye-related ocular symptoms, and who have self-reported use of over the counter ocular wetting agents within the last 120 days.
4. Subjects who meet the following criteria at both screening and Visit 2 (Randomization/Baseline) examinations:

   1. FCS total score ≥ 4 and < 15 in the NEI/Industry Workshop scale, (Appendix 6)
   2. Symptom Severity score of ≥ 40 using the SANDE questionnaire (Appendix 3)
   3. Anesthetized Schirmer test score ≤ 5 mm wetting/5 min
   4. LGCS total score ≥ 5 using the NEI/Industry Workshop scale (where 0=no staining) Note: Subjects must meet all 4 criteria and eligible scores for FCS, Anesthetized Schirmer and LGCS must be in at least one eye and it must be in the same eye at the time of the visit.

Exclusion Criteria:

Subjects meeting any of the following criteria at the Visit 1 (Screening) or Visit 2 (Randomization/Baseline) visits will be excluded:

1. Subjects with any active infectious ocular condition.
2. Subjects who are monocular or have a BCVA, using corrective lenses if necessary, of +1.0 logMAR or worse as assessed by Early Treatment Diabetic Retinopathy Study (ETDRS).
3. Subjects with ocular inflammatory conditions (e.g., conjunctivitis, keratitis, anterior blepharitis, etc.) not related to dry eye syndrome.
4. Subjects with clinical evidence of cicatricial ocular surface disease, such as cicatricial ocular pemphigoid or Stevens Johnson syndrome.
5. Subjects who cannot suspend the use of any topical eye medications (including topical cyclosporine) other than the investigational product during the run-in and the study treatment phase.
6. Subjects who have used Restasis® (topical ophthalmic cyclosporine) or Xiidra® (topical ophthalmic lifitegrast) within 14 days prior to Visit 1.
7. Subjects who in the study eye have fluorescein corneal staining (FCS) Total Score = 15 or a Score = 3 in the superior region per the NEI/Industry Workshop scale or subjects who have FCS with diffuse confluent staining, filaments or frank epithelial defects.
8. Subjects who have active or have had an outbreak of herpetic keratitis within 365 days of Visit 1 or subjects who are on chronic oral antivirals for ocular herpetic disease.
9. Subjects who cannot suspend the use of and abstain from contact lens use from the Screening Visit (Visit 1) to the end of the study (Visit 5).
10. Subjects who have a history of collagen vascular disease, auto immune disease or rheumatic disease other than Primary Sjögren's Syndrome (e.g., Lupus, Rheumatoid Arthritis, etc.).
11. Subjects who have a history of or current Anterior Membrane Dystrophy.
12. Subjects who have had a corneal transplant or similar corneal surgery (DALK, DSEK, DMEK, etc.).
13. Subjects who have used or anticipate use of amiodarone.
14. Subjects who within 30 days prior to Visit 1 alter the dose or anticipate alterations to the dose of the following: tetracyclines, Omega 3's or 6's.
15. Subjects who within 60 days prior to Visit 1 and for the duration of the study alter the dose or anticipate alterations to the dose of the following: anticholinergics, antidepressants, oral contraceptives, isotretinoin, oral systemic corticosteroids, oral systemic immunosuppressive agents.
16. Subjects who within 30 days prior to Visit 1 and for the duration of the study use topical ocular antihistamines, ocular, inhaled or intranasal corticosteroids, topical or oral mast cell stabilizers, oral antihistamines, topical or nasal vasoconstrictors, topical ocular NSAIDs, topical ocular antibiotics or serum tears.
17. Subjects who in the study eye have had cauterization of the punctum or alterations to (insertion or removal) punctal plug(s) within the past 14 days prior to Visit 1. Note: If a punctal plug in place at Visit 2 (Randomization/Baseline) and it is dislodged, the plug should be replaced as soon as possible.
18. Subjects who, in the study eye, have had corneal refractive surgery (LASIK, PRK, RK).
19. Subjects who in the study eye, have a history of any operative procedure on the ocular surface or eyelids within 365 days prior to Visit 1 or with a history of intraocular surgery within 90 days prior to Visit 1.
20. Subjects who are pregnant or suspected to be pregnant and subjects who are breastfeeding or intend to breastfeed. Female subjects of childbearing potential are required to have a negative urine pregnancy test at screening, and must agree to use an acceptable method of contraception from the time of signing informed consent until the end of study visit. Medically acceptable contraception methods include intrauterine device; barrier methods such as diaphragm, condom, cap or sponge, used with a spermicide; or hormonal contraception.
21. Subjects with any physical or mental impairment that would preclude participation and the ability to give informed consent.
22. Subjects who have participated in a device or Investigational drug study or clinical trial within 30 days of Visit 1. Participation in another during this study is excluded for the duration of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Change in Fluorescein Corneal Staining total score | Changes at Week 4 from Baseline
  Mean change from Baseline/Randomization (Visit 2) to Day 28 (Visit 4) in Fluorescein Corneal Staining (FCS) total score [National Eye Institute (NEI)/Industry Workshop 0-15 scale, 0-3 scale in each of 5 regions] in the study eye.

SECONDARY OUTCOMES:
Eye Dryness | Changes at Week 4 from Baseline
  Mean change from Baseline/Randomization (Visit 2) to Day 28 (Visit 4) in Eye Dryness Score (0-100 VAS scale, OU) from Individual Symptom Assessments (Instantaneous)
Mean Scores for Individual Symptom Assessments (Reflective) | Day 28
  Mean Scores for six Individual Symptom Assessments (Reflective) at Day 28 (Visit 4). The individual reflective symptom assessment is assessed in 6 categories (Eye Dryness, Burning/Stinging, Foreign Body Sensation, Eye Discomfort, Eye Pain and Fluctuating Vision). An anchor in the middle at 50 mm representing their symptom severity at the last visit. The 50 mm scale to the left of the anchor located in the center of the scale will measure worsening symptoms (a negative value) and the 50 mm scale to the right of the anchor located in the center of the scale will measure improving symptoms (a positive value). The lower score represents greater severity.
Changes in SANDE-1 to Visit 4 | Changes from Baseline to Day 28.
  Changes in Symptom Assessment in Dry Eye Questionnaires (SANDE) Version 1 global score from Randomization/Baseline (Visit 2) to Day 28 (Visit 4). SANDE Version 1 questionnaire contains two items measuring the frequency and severity of dry eye symptoms. Each item is assessed on a 100 mm visual analog scale from 0 (Rarely for frequency, Very mild for severity) to 100 mm (All the time for frequency, Very Severe for severity), with higher scores representing greater frequency/severity.
Mean Scores SANDE 2 | Day 28
  Mean Scores for Symptom Assessment in Dry Eye Questionnaires (SANDE) Version 2 global scores at day 28 (Visit 4). SANDE Version 2 questionnaire contains two items measuring the frequency and severity of dry eye symptoms.The 50 mm scale to the left of the anchor located in the center of the scale will measure improving symptoms (a negative value) and the 50 mm scale to the right of the anchor located in the center of the scale will measure worsening symptoms (a positive value).
Changes in Individual Symptom Assessments (Instantaneous) | Changes at Baseline to Day 28
  Changes in each of the 5 additional Individual Symptom Assessment (Instantaneous) from Randomization/Baseline (Visit 2) to Day 28 (Visit 4). The individual instantaneous symptom assessment is a questionnaire that uses a 0-100 mm visual analog scale to rate the severity of each ocular symptom for both eyes (OU). There are six categories (Eye Dryness, Burning/Stinging, Foreign Body Sensation, Eye Discomfort, Eye Pain and Fluctuating Vision). The higher score represents more severe symptoms.
Changes in LGCS | Changes at Week 4 from Baseline
  Changes in Lissamine Green Conjunctival Staining (LGCS) from Randomization/Baseline (Visit 2) to Day 28 (Visit 4) in the study eye.
Changes in Anesthetized Schirmer test | Changes at Week 4 from Baseline
  Change in Anesthetized Schirmer test from Randomization/Baseline (Visit 2) to Day 28 (Visit 4) in the study eye.
Changes in Tear Film Break Up Time (TFBUT) | Changes at Week 4 from Baseline
  Changes in tear film break up time (TFBUT) from Randomization/Baseline (Visit 2) to Day 28 (Visit 4) in the study eye
Changes in FCS at Post-Treatment | Baseline to Visit 5 / Day 42
  Changes in Fluorescein Corneal Staining (FCS) from Randomization/Baseline (Visit 2) to the Post-Treatment Follow-Up Visit (day 42) in the study eye. The FCS assessment will be performed for each of the five sections (Central, Inferior, Superior, Temporal, and Nasal) on both eyes (study eye and fellow eye) using the National Eye Institute (NEI)/Industry Workshop scale. The staining in each of the 5 sections of the cornea is evaluated per the NEI score: Grades of 0, 1, 2, and 3 with higher grades representing greater severity.
Changes in SANDE-1 to Visit 5 | Baseline to Visit 5 / Day 42
  Changes in Symptom Assessment in Dry Eye Questionnaires (SANDE) Version 1 global score from Randomization/Baseline (Visit 2) to the Post Treatment Follow-up visit (Day 42). SANDE Version 1 questionnaire contains two items measuring the frequency and severity of dry eye symptoms. Each item is assessed on a 100 mm visual analog scale from 0 (Rarely for frequency, Very mild for severity) to 100 mm (All the time for frequency, Very Severe for severity), with higher scores representing greater frequency/severity.
Changes in Individual Symptom Assessments (Instantaneous) from Baseline Visit 5 | Baseline to Visit 5
  Changes in six Individual Symptoms (Instantaneous) from Randomization/Baseline (Visit 2) to the Post-Treatment Follow-up Visit (Day 42). The individual instantaneous symptom assessment is a questionnaire that uses a 0-100 mm visual analog scale to rate the severity of each ocular symptom. There are six categories (Eye Dryness, Burning/Stinging, Foreign Body Sensation, Eye Discomfort, Eye Pain and Fluctuating Vision). The higher score represents more severe symptoms.
Mean Scores for SANDE-2 | Visit 5 / Day 42
  Mean Scores for Symptom Assessment in Dry Eye Questionnaires (SANDE) Version 2 global score at the Post-Treatment Follow-Up Visit (Day 42). SANDE Version 2 questionnaire contains two items measuring the frequency and severity of dry eye symptoms.The 50 mm scale to the left of the anchor located in the center of the scale will measure improving symptoms (a negative value) and the 50 mm scale to the right of the anchor located in the center of the scale will measure worsening symptoms (a positive value).
Mean Scores for six Individual Symptom Assessments (Reflective) | Visit 5 / Day 42
  Mean Scores for six Individual Symptom Assessments (Reflective) at the Post-Treatment Follow-Up Visit (Day 42). The individual reflective symptom assessment is assessed in 6 categories (Eye Dryness, Burning/Stinging, Foreign Body Sensation, Eye Discomfort, Eye Pain and Fluctuating Vision). The 50 mm scale to the left of the anchor located in the center of the scale will measure worsening symptoms (a negative value) and the 50 mm scale to the right of the anchor located in the center of the scale will measure improving symptoms (a positive value).
Changes in FCS | Baseline to Day 28
  Mean change from Baseline/Randomization (Visit 2) to Day 28 (Visit 4) in Fluorescein Corneal Staining (FCS) total score [National Eye Institute (NEI)/Industry Workshop 0-15 scale, 0-3 scale in each of 5 regions] in the qualifying fellow eye.
Changes in LCGS Anesthetized Schirmer test, TFBUT | Baseline to Day 28
  Changes in Lissamine Green Conjunctival Staining (LCGS) Anesthetized Schirmer test, tear film break up time (TFBUT) from Randomization/Baseline (Visit 2) to Day 28 (Visit 4) in the qualifying fellow eye.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Odrich, MD, Study Director — TearSolutions, Inc.
Locations (35):
- United States (35):
  - University of Alabama Eye Center, Birmingham, Alabama
  - Doctor My Eyes / Stephen Cohen, OD, PC, Scottsdale, Arizona
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - Milton M. Hom, OD FAAO FACAA (Sc), Azusa, California
  - University of California, Berkeley, School of Optometry, Berkeley, California
  - Orange County Ophthalmology, Garden Grove, California
  - Lugene Eye Institute, Glendale, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - University of Colorado Department of Ophthalmology, Aurora, Colorado
  - Corneal Consultants of Colorado, Littleton, Colorado
  - Bruce A. Segal, MD PA Private Practice, Delray Beach, Florida
  - Bowden Eye & Associates, Jacksonville, Florida
  - International Eye Associates, PA, Ormond Beach, Florida
  - Perez Eye Center, Tampa, Florida
  - Eye Consultants of Atlanta, Atlanta, Georgia
  - Chicago Cornea Consultants, Ltd., Hoffman Estates, Illinois
  - Midwest Cornea Associates, LLC, Indianapolis, Indiana
  - The Eye Care Institute, Louisville, Kentucky
  - Clinical Eye Research of Boston, Winchester, Massachusetts
  - Minnesota Eye Consultants, P.A., Bloomington, Minnesota
  - Tauber Eye Center, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Cornea Consultants of Albany, Slingerlands, New York
  - Cornerstone Eye Care, PA, High Point, North Carolina
  - Bergstrom Eye Research, Fargo, North Dakota
  - Abrams Eye Center, Cleveland, Ohio
  - Ophthalmic Surgeons & Consultants of Ohio; The Eye Center of Columbus, Columbus, Ohio
  - University of Pennsylvania Scheie Eye Institute, Philadelphia, Pennsylvania
  - Black Hills Eye Institute, Rapid City, South Dakota
  - UTHSC Department of Ophthalmology, Memphis, Tennessee
  - The Eye Clinic of Texas, an affiliate of Houston Eye Associates, League City, Texas
  - University of Virginia University Eye Center, Charlottesville, Virginia
  - Virginia Eye Consultants, Norfolk, Virginia
  - Vistar Eye Center, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No